CLINICAL TRIAL: NCT01728415
Title: Effects of High-intensity Interval Training in Patients in Hemodialysis
Acronym: OsloExDia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Responsible Party: Principal Investigator, Birgitta Blakstad Nilsson, PhD, The Oslo ExDia-study, Oslo University Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/1459; 126/12-303.0 (Other Grant/Funding Number: The Norwegian Fund for Post-Graduate Training in Physiotherapy)
Record Dates: First submitted 2012-11-13; First posted 2012-11-19 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Renal Disease
Keywords: Exercise; Hemodialysis; Physical therapy; high-intensity
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A: Exercise (Experimental): High intensity interval exercise training (3 x 3 minutes of intensity abow 85% og Heart rate peak)
  Interventions: Other: exercise
- B: Execise (Active Comparator): Moderate continuous exercise training
  Interventions: Other: exercise
- C: Controll (No Intervention): Usual care without exercise training

INTERVENTIONS:
Other: exercise — Group A: high intensity exercise training Group B: moderate intensity exercise training C: Control group
  Arms: A: Exercise; B: Execise

SUMMARY:
The purpose of this study is to evaluate the effects of high intensity interval training compared to moderate exercise training and a control group on exercise capacity and quality of life in patients with end stage renal disease on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients on hemodialysis ≥ 3 months

Exclusion Criteria:

* Acute infection
* Systolic BP>180 mmHG or diabolic BP>105 mmHG
* Unstable angina pectoris
* Serious rhythm disturbances
* Hyperkalemic (> 6 mmol/L),
* Unstable diabetes mellitus
* Wheelchair
* Dialyses access on lower extremities
* Haemoglobin < 9 g/dl

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-12 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen uptake | baseline, 16 weeks
  Canges from baseline in peak oxygen uptake at 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Postboks 4950 Nydalen, Norway

REFERENCES:
- [Derived] Nilsson BB, Bunaes-Naess H, Edvardsen E, Stenehjem AE. High-intensity interval training in haemodialysis patients: a pilot randomised controlled trial. BMJ Open Sport Exerc Med. 2019 Nov 10;5(1):e000617. doi: 10.1136/bmjsem-2019-000617. eCollection 2019. PMID 31798950